CLINICAL TRIAL: NCT00113490
Title: A Phase 1/2 Study to Evaluate the Safety, Tolerability, and Immunogenicity of MEDI-524, a Humanized Enhanced Potency Monoclonal Antibody Against Respiratory Syncytial Virus (RSV), After Dosing for a Second Season in Children Who Previously Received MEDI-524 in Protocol MI-CP104
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of Motavizumab (MEDI-524) After Dosing for a Second Season in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP118
Record Dates: First submitted 2005-06-08; First posted 2005-06-09 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-04

CONDITIONS: Motavizumab Administration for a Second Season for RSV Prophylaxis
Keywords: motavizumab, palivizumab, synagis; Rezield, MEDI-524
MeSH Terms: interventions — motavizumab; Palivizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- motavizumab (MEDI-524) 15 mg/kg (Experimental): A single IM injection every 30 days beginning at Day 0 for a total of 4-5 injections determined by when in the RSV season a child was enrolled.
  Interventions: Biological: motavizumab (MEDI-524)
- palivizumab 15 mg/kg (Active Comparator): A single IM injection every 30 days beginning at Day 0 for a total of 4-5 injections determined by when in the RSV season a child was enrolled.
  Interventions: Biological: palivizumab 15 mg/kg

INTERVENTIONS:
Biological: motavizumab (MEDI-524) — Patients will receive 15 mg/kg MEDI-524 administered IM every 30 days for a total of 4-5 injections.
  Other Names: motavizumab; Rezield
  Arms: motavizumab (MEDI-524) 15 mg/kg
Biological: palivizumab 15 mg/kg — Patients will receive 15 mg/kg palivizumab administered IM every 30 days for a total of 4-5 injections.
  Other Names: synagis
  Arms: palivizumab 15 mg/kg

SUMMARY:
The primary objective of this study was to determine the effect on immune reactivity to motavizumab (MEDI-524) of monthly intramuscular (IM) doses of motavizumab (MEDI-524) administered for a second season in children.

DETAILED DESCRIPTION:
This was a Phase 1/2, randomized, double-blind study in which motavizumab (MEDI-524) or palivizumab was administered to children who previously participated in MI-CP104. Children who received at least 3 doses of motavizumab in MI-CP104 were eligible for enrollment. Subjects were randomized 1:1 to receive motavizumab or palivizumab at 15 mg/kg by IM injection every 30 days for a total of 4-5 injections during the 2004-05 RSV season subsequent to the season in which they were participants of MI-CP104. All subjects were evaluated prior to and 30 minutes after each injection of study drug with 2 follow-up evaluations, one at 30 days and the other at 90-120 days after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in MI-CP104 and received at least 3 injections of MEDI-524 in MI-CP104
* The child must be less than or equal to 24 months of age at time of entry into the study (child must be entered on or before their 24-month birthday)
* The child must be able to complete the follow-up visits through 3-4 months after last dose (total length of participation of 6-8 months)
* Written informed consent obtained from the patient's parent(s) or legal guardian

Exclusion Criteria:

* Currently hospitalized
* Receiving chronic oxygen therapy or mechanical ventilation at the time of study entry (including continuous positive airway pressure [CPAP])
* Evidence of infection with hepatitis A, B, or C virus
* Known renal impairment, hepatic dysfunction, chronic seizure disorder, or immunodeficiency or HIV infection
* Suspected serious allergic or immune mediated events with prior receipt of MEDI-524
* Acute illness or progressive clinical disorder
* Active infection, including acute respiratory syncytial virus (RSV) infection at the time of enrollment
* Previous reaction to IGIV, blood products, or other foreign proteins
* Have ever received palivizumab
* Received within the past 120 days or currently receiving immunoglobulin products (such as RSV-IGIV [RespiGam(R)], IVIG), or any investigational agents (except MEDI-524)
* Currently participating in any investigational study

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2005-05; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Pamela Griffin, M.D., Study Director — MedImmune LLC
Locations (6):
- Brazil (2):
  - Pontificia Universidade Catolica Do Rio Grande, Porto Alegre
  - Hospital Das Clinicas Da Faculdade, Ribeirão Preto
- Chile (4):
  - Hospital Clinico De La Pointificia Universidad, Santiago
  - Hospital Clinico de la Universidad de Chile, Santiago
  - Hospital Dr. Sotero Del Rio, Santiago
  - Hospital San Jose, Santiago

REFERENCES:
- [Result] Abarca K, Jung E, Fernandez P, Zhao L, Harris B, Connor EM, Losonsky GA; Motavizumab Study Group. Safety, tolerability, pharmacokinetics, and immunogenicity of motavizumab, a humanized, enhanced-potency monoclonal antibody for the prevention of respiratory syncytial virus infection in at-risk children. Pediatr Infect Dis J. 2009 Apr;28(4):267-72. doi: 10.1097/INF.0b013e31818ffd03. PMID 19258920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children who received at least 3 doses of motavizumab in Study MI-CP104 during the 2004-2005 RSV season were eligible for enrollment in this study. It was anticipated that approximately 150 children would be enrolled.
Pre-assignment Details: Motavizumab or palivizumab was administered to children, using a 1:1 randomization, at 15 mg/kg of study drug by IM injection every 30 days, for a total of 4-5 doses (determined by when in the RSV season a child was enrolled) during the 2005-2006 RSV season.
Groups:
- Motavizumab (MEDI-524) 15 mg/kg; Palivizumab 15 mg/kg: A single intramuscular injection every 30 days for a total of 4-5 injections determined by when in the RSV season a child was enrolled.
Period: Overall Study
Arm/Group | Motavizumab (MEDI-524) 15 mg/kg | Palivizumab 15 mg/kg
Started | 66 | 70
Completed | 64 | 67
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motavizumab (MEDI-524) 15 mg/kg | Palivizumab 15 mg/kg | Total
Number analyzed (Participants) | 66 | 70 | 136
Age Continuous [Mean (Standard Deviation); unit: Months] | 13.25 (3.13) | 13.59 (2.89) | 13.43 (3.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 32 | 55
  Male | 43 | 38 | 81
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 61 | 62 | 123
  White/Non-Hispanic | 5 | 6 | 11
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Exhibiting Anti-motavizumab Antibodies
Description: Serum for measurement of anti-motavizumab antibodies was collected prior to the first, second and, if applicable, fifth doses of study drug, and at the 2 follow-up visits 30 and 90-120 days post final dose.
Time Frame: Day 0 through 120 days post final dose
Population: All subjects who received any study drug were included in all summaries of immunogenicity. Day 0 n=66 mota, n=70 pali; Day 25-30 n=65 mota, n=69 pali; Day 120 n=64 mota, n=67 pali; 30 days post final dose n=65 mota, n=67 pali; 90-120 days post final dose n=64 mota, n=67 pali; at any time n=66 mota, n=70 pali.
Measure: Number; unit: participants
Arm/Group | Motavizumab (MEDI-524) 15 mg/kg | Palivizumab 15 mg/kg
Number analyzed (Participants) | 66 | 70
participants
  Day 0 | 2 | 3
  Day 25-30 | 0 | 3
  Day 120 | 0 | 6
  30 Days Post Final Dose | 0 | 9
  90-120 Days Post Final Dose | 0 | 10
  At any time | 2 | 12

2. Secondary Outcome: Number of Subjects Reporting Adverse Events (AEs)
Description: Assessments of adverse events (including SAEs) were made by clinical investigators according to the protocol.
Time Frame: Day 0 through 30 days post final dose
Population: All subjects who received any study drug were included in all summaries of safety.
Measure: Number; unit: participants
Arm/Group | Motavizumab (MEDI-524) 15 mg/kg | Palivizumab 15 mg/kg
Number analyzed (Participants) | 66 | 70
participants | 56 | 62

3. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: Assessments of SAEs were made by clinical investigators according to the protocol.
Time Frame: Day 0 through 30 days post final dose
Population: All subjects who received any study drug were included in all summaries of safety.
Measure: Number; unit: participants
Arm/Group | Motavizumab (MEDI-524) 15 mg/kg | Palivizumab 15 mg/kg
Number analyzed (Participants) | 66 | 70
participants | 4 | 1

4. Secondary Outcome: Number of Subjects With Increased Toxicity Grade From Baseline as Determined by Laboratory Evaluations
Description: Serum chemistry and hematology parameters were measured at baseline, on Days 25-30 and 120, 30 days post the final dose, and at premature discontinuation.
Time Frame: Day 0 through 30 days post final dose
Population: All subjects who received any study drug were included in all summaries of safety.
Measure: Number; unit: participants
Arm/Group | Motavizumab (MEDI-524) 15 mg/kg | Palivizumab 15 mg/kg
Number analyzed (Participants) | 66 | 70
participants
  ALT Increased | 1 | 0
  Blood Urea Nitrogen Increased | 0 | 4
  Anemia | 3 | 3
  Eosinophil Count Increased | 0 | 2
  Neutropenia | 0 | 2
  AST increased | 0 | 2
  Hemoglobin Decreased | 1 | 0
  Eosinophilia | 3 | 4

5. Secondary Outcome: Motavizumab Serum Concentrations at Each Data Collection Visit
Description: Mean serum concentration.
Time Frame: Prior to dosing on Day 0, Day 30, Day 120, and at 30 and 90-120 days post final dose
Population: All subjects who received any study drug were included in all summaries. Day 0 n= 66; Day 25-30 n=65; Day 120 n=63; 30 days post final dose n=63; 90-120 days post final dose n=62
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Motavizumab (MEDI-524) 15 mg/kg
Number analyzed (Participants) | 66
ug/mL
  Day 0 | 1.536 (6.192)
  Day 25-30 | 54.59 (16.05)
  Day 120 | 86.21 (23.79)
  30 Days Post Final Dose | 76.03 (27.13)
  90-120 Days Post Final Dose | 12.2 (6.260)

ADVERSE EVENTS:
Time Frame: Day 0 through 30 days post final dose.
Arm/Group | Motavizumab (MEDI-524) 15 mg/kg | Palivizumab 15 mg/kg
Serious Adverse Events (participants affected / at risk) | 4/66 | 1/70
Other Adverse Events (participants affected / at risk) | 56/66 | 62/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motavizumab (MEDI-524) 15 mg/kg (N=66) | Palivizumab 15 mg/kg (N=70)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
PNEUMONITIS CHEMICAL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motavizumab (MEDI-524) 15 mg/kg (N=66) | Palivizumab 15 mg/kg (N=70)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
BLOOD UREA INCREASED (Investigations) | 0 (0) | 4 (4)
BRONCHITIS (Infections and infestations) | 21 (33) | 19 (38)
CANDIDA NAPPY RASH (Infections and infestations) | 3 (3) | 2 (2)
CONJUNCTIVITIS (Eye disorders) | 4 (4) | 4 (4)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
DIARRHOEA (Gastrointestinal disorders) | 11 (12) | 10 (13)
EOSINOPHILIA (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
IMMUNISATION REACTION (Immune system disorders) | 2 (2) | 4 (4)
INJECTION SITE ERYTHEMA (General disorders) | 10 (16) | 8 (10)
LARYNGITIS (Infections and infestations) | 3 (4) | 4 (4)
NASOPHARYNGITIS (Infections and infestations) | 29 (38) | 29 (44)
OTITIS MEDIA (Infections and infestations) | 1 (1) | 3 (3)
OTITIS MEDIA ACUTE (Infections and infestations) | 4 (5) | 3 (3)
PHARYNGITIS (Infections and infestations) | 6 (6) | 8 (10)
PNEUMONIA (Infections and infestations) | 2 (2) | 3 (3)
PRURIGO (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
PYREXIA (General disorders) | 2 (2) | 4 (4)
RHINITIS (Infections and infestations) | 6 (6) | 4 (6)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
TONSILLITIS (Infections and infestations) | 4 (6) | 5 (5)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 4 (5)
VARICELLA (Infections and infestations) | 3 (3) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 14 (19) | 16 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.The PIs also agree for data to be presented first as a joint, multi-center publication.